CLINICAL TRIAL: NCT02752776
Title: An Open-label, Prospective, Non-randomized, Multicenter Study to Evaluate Clear Skin Effect on Health Related Quality of Life Outcomes at 16 and 52 Weeks in Patients With Moderate to Severe Plaque Psoriasis Treated With Secukinumab 300 mg s.c. With or Without Previous Exposure to Systemic Therapy.
Brief Title: A Study to Evaluate Clear Skin Effect on Quality of Life in Patients With Plaque Psoriasis.
Acronym: PROSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAIN457A3401; 2015-003701-42 (EudraCT Number)
Record Dates: First submitted 2016-02-10; First posted 2016-04-27 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-08

CONDITIONS: Plaque Psoriasis
Keywords: secukinumab; AIN457; Moderate to severe plaque psoriasis; immune-mediated systemic disease; scaly patches; papules; plaques; itching
MeSH Terms: conditions — Plaque, Amyloid; Pruritus | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Secukinumab (Experimental): All patients are received s.c. injections of secukinumab 300 mg at Week 0, 1, 2 and 3 during the first 4 weeks followed by monthly maintenance dosing of 300 mg secukinumab starting at Week 4 until Week 48. Consideration was given to discontinuing treatment in patients who showed no response up to 16 weeks of treatment (e.g. patients who did not achieve a PASI 50 response). If discontinued, patients completed the end of study visit assessments. Some patients with an initially partial response (e.g. patients who achieved a PASI 50 response but not a PASI 75 response) subsequently improved with continued treatment beyond 16 weeks.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Secukinumab was used as commercially available PFS of 150 mg. Patients received PFS at the site and were instructed to administer Secukinumab as needed (300 mg each application).
  Other Names: AIN457

SUMMARY:
Study of effects of secukinumab 300 mg s.c. on quality of life (QoL) in psoriasis in patients with or without prior exposure to systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged at least 18 years at time of Screening.
* Moderate to severe plaque-type psoriasis diagnosed for at least 3 months prior to Screening and candidate for systemic therapy.
* Other protocol defined inclusion criteria may apply. Please refer to the protocol.

Exclusion Criteria:

* Forms of psoriasis other than moderate to severe plaque-type psoriasis, e.g. drug-induced psoriasis at Screening.
* Patients with previous treatment with any agent targeting interleukin (IL)-17 directly or IL-17 receptor A (e.g. secukinumab, ixekizumab, or brodalumab).
* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless they use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1660 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (190):
- Belgium (4):
  - Novartis Investigative Site, Geel, BEL
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Seraing
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Varna
- Czechia (3):
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- France (33):
  - Novartis Investigative Site, Le Mans, Cedex 09
  - Novartis Investigative Site, Toulon, Val De Marne
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Argenteuil
  - Novartis Investigative Site, Auxerre
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Boulogne-sur-Mer
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Cannes
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Martigues
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Pringy
  - Novartis Investigative Site, Quimper
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Mandé
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Valence
  - Novartis Investigative Site, Valenciennes
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (34):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Andernach
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bramsche
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Friedrichshafen
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Ibbenbueren
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Ludwigshafen am Rhein
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Pommelsbrunn
  - Novartis Investigative Site, Quedlinburg
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Simmern
  - Novartis Investigative Site, Vechta
  - Novartis Investigative Site, Wiesbaden
- Greece (3):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Pátrai
- Israel (5):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
- Italy (7):
  - Novartis Investigative Site, Arezzo, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, San Donato Milanese, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Varese, VA
- Latvia (5):
  - Novartis Investigative Site, Daugavpils, LVA
  - Novartis Investigative Site, Jelgava, LVA
  - Novartis Investigative Site, Riga, LVA
  - Novartis Investigative Site, Ventspils, LVA
  - Novartis Investigative Site, Riga
- Lithuania (4):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Klaipėda, LTU
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Vilnius
- Poland (11):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Ossy
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (3):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Nova de Gaia
- Romania (4):
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Iași
- Slovakia (7):
  - Novartis Investigative Site, Malacky, Slovak Republic
  - Novartis Investigative Site, Bardejov, SVK
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Svidník
  - Novartis Investigative Site, Žilina
- Spain (40):
  - Novartis Investigative Site, Ferrol, A Coruna
  - Novartis Investigative Site, Vitoria-Gasteiz, Alava
  - Novartis Investigative Site, Elda, Alicante
  - Novartis Investigative Site, Almería, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Barakaldo, Basque Country
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Jerez de la Frontera, Cadiz
  - Novartis Investigative Site, Ávila, Castille and León
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Albacete, Castille-La Mancha
  - Novartis Investigative Site, Guadalajara, Castille-La Mancha
  - Novartis Investigative Site, Toledo, Castille-La Mancha
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Terrassa, Catalonia
  - Novartis Investigative Site, Zamora, Espana
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Ourense, Galicia
  - Novartis Investigative Site, Alcalá de Henares, Madrid
  - Novartis Investigative Site, Aranjuez, Madrid
  - Novartis Investigative Site, Fuenlabrada, Madrid
  - Novartis Investigative Site, Getafe, Madrid
  - Novartis Investigative Site, Leganés, Madrid
  - Novartis Investigative Site, Torrejón de Ardoz, Madrid
  - Novartis Investigative Site, Móstoles, Madrid, Communidad de
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Breña Alta, Santa Cruz De Tenerife
  - Novartis Investigative Site, Talavera de la Reina, Toledo
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Burgos
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, Granollers
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Zaragoza
- United Kingdom (21):
  - Novartis Investigative Site, Penzance, Cornwall
  - Novartis Investigative Site, Harlow, Essex
  - Novartis Investigative Site, Rothwell, GBR
  - Novartis Investigative Site, Burbage, Leicester
  - Novartis Investigative Site, Harrow, Middlesex
  - Novartis Investigative Site, Bury Saint Edmonds, Suffolk
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Chippenham
  - Novartis Investigative Site, Devon
  - Novartis Investigative Site, Durham
  - Novartis Investigative Site, East Sussex
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Lancaster
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Middlesex
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Stoke-on-Trent
  - Novartis Investigative Site, Watford
  - Novartis Investigative Site, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
Supporting Information: Study Protocol, SAP
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] da Silva N, Sommer R, Ortmann CE, Jagiello P, Bachhuber T, Augustin M. Secukinumab effects on disease burden, patient needs and benefits, and treatment satisfaction in patients with plaque psoriasis across European regions: patient perspective data from the PROSE study. J Eur Acad Dermatol Venereol. 2021 Nov;35(11):2241-2249. doi: 10.1111/jdv.17525. Epub 2021 Jul 31. PMID 34273904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1660 participants were treated and included in the Safety set.
Pre-assignment Details: A total of 1858 patients were screened in this study.
Groups:
- Subpopulation A (Naive): Participants who were naïve to any systemic treatment, e.g. participants failing or intolerant to previous topical treatment, including narrow band UVB, but never exposed to any systemic treatment, with or without contraindications to the use of conventional systemic treatment and in a need of a first systemic treatment.
- Subpopulation B (Non-biologic): Participants who have been previously exposed to at least one conventional systemic therapy; either because of failure or intolerance to their previous conventional systemic treatment, they were in a need of a first biologic systemic treatment.
- Subpopulation C (Biologic): Participants who have been previously exposed to at least one biologic systemic therapy; either because of failure or intolerance to their previous biologic systemic treatment, they were in a need of a different biologic systemic treatment.
Period: Overall Study
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic)
Started | 663 | 673 | 324
Completed | 611 | 597 | 276
Not Completed | 52 | 76 | 48
Not completed — Adverse Event | 15 | 23 | 11
Not completed — Lack of Efficacy | 2 | 6 | 14
Not completed — Lost to Follow-up | 11 | 12 | 4
Not completed — Non-compliance with study treatment | 0 | 0 | 1
Not completed — Physician Decision | 2 | 6 | 2
Not completed — Pregnancy | 1 | 6 | 3
Not completed — Protocol Violation | 10 | 13 | 6
Not completed — Subject/guardian decision | 8 | 6 | 4
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety set: The Safety set included all patients who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | Total
Number analyzed (Participants) | 663 | 673 | 324 | 1660
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (14.03) | 44.4 (13.67) | 47.4 (12.89) | 44.5 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 222 | 107 | 553
  Male | 439 | 451 | 217 | 1107
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 626 | 642 | 307 | 1575
  Black | 3 | 2 | 0 | 5
  Asian | 12 | 6 | 2 | 20
  Other | 22 | 23 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Dermatology Life Quality Index 0/1 (DLQI 0/1) Response at Week 16
Description: The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne and viral worts. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment.
Time Frame: 16 weeks
Population: Full Analysis set: The Full Analysis set included all patients who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Participants: Participants from all 3 subpopulations: Subpopulation A B & C combined
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
Number analyzed (Participants) | 662 | 673 | 324 | 1659
Percentage of participants | 74.7 [71.2 to 78.0] | 71.3 [67.7 to 74.7] | 61.7 [56.1 to 67.0] | 70.8 [68.5 to 73.0]

2. Secondary Outcome: Percentage of Participants With a Dermatology Life Quality Index 0/1 (DLQI 0/1) Response at Week 52
Description: as for outcome 1
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
Number analyzed (Participants) | 662 | 673 | 324 | 1659
Percentage of participants | 75.3 [71.7 to 78.5] | 73.3 [69.8 to 76.6] | 62.0 [56.5 to 67.3] | 71.9 [69.6 to 74.0]

3. Secondary Outcome: Percentage of Participants in Each DLQI Score Category at Week 16 and Week 52
Description: as for outcome 1
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
Number analyzed (Participants) | 662 | 673 | 324 | 1659
Percentage of participants
  Wk 16: DLQI cat. score: 2-5: number analyzed (Participants) | 649 | 666 | 321 | 1636
  Wk 16: DLQI cat. score: 2-5 | 18.3 [15.5 to 21.6] | 19.1 [16.2 to 22.3] | 21.2 [16.9 to 26.2] | 19.2 [17.3 to 21.2]
  Wk 16: DLQI cat. score: 6-10: number analyzed (Participants) | 649 | 666 | 321 | 1636
  Wk 16: DLQI cat. score: 6-10 | 5.7 [4.1 to 7.8] | 6.3 [4.6 to 8.5] | 9.3 [6.5 to 13.2] | 6.7 [5.5 to 8.0]
  Wk 16: DLQI cat. score: 11-20: number analyzed (Participants) | 649 | 666 | 321 | 1636
  Wk 16: DLQI cat. score: 11-20 | 1.2 [0.6 to 2.5] | 2.9 [1.8 to 4.5] | 5.3 [3.2 to 8.5] | 2.7 [2.0 to 3.6]
  Wk 16:DLQI cat. score: 21-30: number analyzed (Participants) | 649 | 666 | 321 | 1636
  Wk 16:DLQI cat. score: 21-30 | 0.0 [0.0 to 0.7] | 0.5 [0.1 to 1.4] | 2.5 [1.2 to 5.0] | 0.7 [0.4 to 1.2]
  Wk 52: DLQI cat. score: 2-5: number analyzed (Participants) | 655 | 671 | 324 | 1650
  Wk 52: DLQI cat. score: 2-5 | 17.9 [15.0 to 21.1] | 14.0 [11.5 to 16.9] | 18.2 [14.2 to 23.0] | 16.4 [14.6 to 18.3]
  Wk 52: DLQI cat. score: 6-10: number analyzed (Participants) | 655 | 671 | 324 | 1650
  Wk 52: DLQI cat. score: 6-10 | 4.7 [3.3 to 6.7] | 7.2 [5.4 to 9.4] | 9.6 [6.7 to 13.4] | 6.7 [5.5 to 8.0]
  Wk 52:DLQI cat. score: 11-20: number analyzed (Participants) | 655 | 671 | 324 | 1650
  Wk 52:DLQI cat. score: 11-20 | 1.8 [1.0 to 3.3] | 4.0 [2.7 to 5.9] | 8.3 [5.7 to 12.0] | 4.0 [3.1 to 5.1]
  Wk 52:DLQI cat. score: 21-30: number analyzed (Participants) | 655 | 671 | 324 | 1650
  Wk 52:DLQI cat. score: 21-30 | 0.3 [0.1 to 1.2] | 1.5 [0.8 to 2.8] | 1.9 [0.8 to 4.2] | 1.1 [0.7 to 1.8]

4. Secondary Outcome: Percentage of Participants With PASI 50, PASI 75, PASI 90, PASI 100 or IGA Mod 2011 0/1 Response at Week 16 and 52
Description: PASI is a combined assessment of lesion severity & affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs); each area is scored by itself & scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), & severity is estimated by clinical signs, erythema, induration & desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 50, 75, 90 & 100 were defined as participants achieving ≥ 50%, 75%, 90% or 100% improvement from baseline. The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
Time Frame: Week 16, Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
Number analyzed (Participants) | 662 | 673 | 324 | 1659
Percentage of participants
  Wk 16: PASI 50: number analyzed (Participants) | 658 | 670 | 323 | 1651
  Wk 16: PASI 50 | 97.7 [96.2 to 98.7] | 97.5 [95.9 to 98.5] | 95.0 [91.9 to 97.2] | 97.1 [96.1 to 97.8]
  Wk 16: PASI 75: number analyzed (Participants) | 658 | 670 | 323 | 1651
  Wk 16: PASI 75 | 94.4 [92.3 to 96.0] | 92.8 [90.5 to 94.7] | 85.4 [81.0 to 89.1] | 92.0 [90.6 to 93.3]
  Wk 16: PASI 90: number analyzed (Participants) | 658 | 670 | 323 | 1651
  Wk 16: PASI 90 | 82.4 [79.2 to 85.2] | 78.8 [75.5 to 81.8] | 69.0 [63.6 to 74.0] | 78.3 [76.2 to 80.3]
  Wk 16: PASI 100: number analyzed (Participants) | 658 | 670 | 323 | 1651
  Wk 16: PASI 100 | 47.3 [43.4 to 51.2] | 38.8 [35.1 to 42.6] | 33.4 [28.4 to 38.9] | 41.1 [38.7 to 43.6]
  Wk 16: IGA 0/1: number analyzed (Participants) | 658 | 671 | 323 | 1652
  Wk 16: IGA 0/1 | 87.4 [84.5 to 89.8] | 84.9 [82.0 to 87.5] | 76.2 [71.1 to 80.7] | 84.2 [82.3 to 85.9]
  Wk 52: PASI 50 | 97.9 [96.4 to 98.9] | 96.3 [94.5 to 97.6] | 92.9 [89.4 to 95.5] | 96.3 [95.2 to 97.1]
  Wk 52: PASI 75 | 94.4 [92.3 to 96.0] | 89.7 [87.1 to 91.9] | 83.3 [78.7 to 87.2] | 90.4 [88.8 to 91.7]
  Wk 52: PASI 90 | 80.8 [77.6 to 83.7] | 75.5 [72.0 to 78.7] | 63.9 [58.4 to 69.1] | 75.3 [73.2 to 77.4]
  Wk 52: PASI 100 | 56.9 [53.1 to 60.8] | 45.5 [41.7 to 49.3] | 37.0 [31.8 to 42.6] | 48.4 [46.0 to 50.8]
  Wk 52: IGA 0/1 | 86.4 [83.5 to 88.9] | 79.9 [76.7 to 82.9] | 71.3 [66.0 to 76.1] | 80.8 [78.8 to 82.7]

5. Secondary Outcome: Absolute Change From Baseline in EQ-5D-5L Crosswalk Index at Week 16 and Week 52
Description: The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort & anxiety/depression. The 5 dimensions have 5 response levels scored from 1 (best) to 5 (worst). The first 3 dimensions have the response levels lasting from no problems, slight problems, moderate problems, severe problems to unable; the last 2 dimensions have the 5 response levels lasting from no, slight, moderate, severe to extreme. From these 5 dimensions the Crosswalk-index is calculated by concatenating the responses & choosing the corresponding country specific index value from the EQ-5D-5L_Crosswalk_Index_Value_Calculator.v2 excel file (https://euroqol.org/eq-5d-instruments/eq-5d-5labout/valuation-standard-value-sets/crosswalk-index-value-calculator/). This calculated participant-level index scores from -0.654 (worst health) to 1.0 (best health).
Time Frame: Week 16, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
Number analyzed (Participants) | 662 | 673 | 324 | 1659
scores on a scale
  Week 16: number analyzed (Participants) | 643 | 656 | 314 | 1613
  Week 16 | 0.217 (0.2294) | 0.201 (0.2277) | 0.235 (0.2602) | 0.214 (0.2352)
  Week 52: number analyzed (Participants) | 647 | 659 | 317 | 1623
  Week 52 | 0.221 (0.2353) | 0.193 (0.2360) | 0.226 (0.2596) | 0.211 (0.2408)

6. Secondary Outcome: Absolute Change From Baseline in EQ-5D-5L Visual Analogue Scale (VAS) at Week 16 and Week 52
Description: A visual analogue scale (VAS) was used within the EQ-5D. This scale recorded the respondent's self-rated health on a vertical 20-cm VAS where the endpoints were labeled "best imaginable health state" and "worst imaginable health state." This resulted in a numeric value set ranging from 0 (="worst imaginable health state") up to 100 (="best imaginable health state").
Time Frame: Week 16, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
Number analyzed (Participants) | 662 | 673 | 324 | 1659
scores on a scale
  Week 16: number analyzed (Participants) | 644 | 656 | 314 | 1614
  Week 16 | 19.7 (24.36) | 21.4 (25.66) | 18.7 (26.66) | 20.2 (25.36)
  Week 52: number analyzed (Participants) | 647 | 659 | 317 | 1623
  Week 52 | 21.7 (24.11) | 22.6 (25.47) | 19.5 (25.14) | 21.7 (24.88)

7. Secondary Outcome: Absolute Change From Baseline in HAQ-DI at Week 16 and Week 52
Description: The HAQ-DI (Health Assessment Questionnaire - Disability Index) assesses a patient's level of functional ability & includes questions on fine movements of the upper extremity, locomotor activities of the lower extremity & activities that involve both upper & lower extremities. There are 20 items in 8 categories of functioning including dressing & grooming, arising, eating, walking, hygiene, reach, grip & usual activities. The stem of each item asks over the past week, "Are you able to..." perform a particular task. Each item is scored on a 4-point scale from 0 to 3, representing normal, no difficulty (0), some difficulty (1), much difficulty (2) & unable to do (3). The HAQ-DI also includes questions about the use of 'aids or devices' & aid from other people to supplement the answers given to the 20 items. Total scores were calculated by averaging all scores and ranging from 0 (best) to 3 (worst). Subtracting the baseline value from the week 16 or 52 values results in the change.
Time Frame: Week 16 and Week 52
Population: Full Analysis set - subset of patients with psoriatic arthritis at baseline: The Full Analysis set included all patients who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
Number analyzed (Participants) | 44 | 117 | 90 | 251
scores on a scale
  Week 16: number analyzed (Participants) | 43 | 109 | 87 | 239
  Week 16 | -0.7 (0.97) | -0.5 (0.83) | -0.3 (0.85) | -0.5 (0.87)
  Week 52: number analyzed (Participants) | 44 | 110 | 88 | 242
  Week 52 | -0.7 (0.90) | -0.5 (0.90) | -0.4 (0.85) | -0.5 (0.88)

8. Secondary Outcome: Absolute Change From Baseline in Numeric Rating Scale (NRS) at Week 16 and Week 52
Description: Selfadministered 11-point numeric rating scales (NRS, 0-10) were used to evaluate the patients' assessment of their current pain, itching & scaling. Respondents answered the following questions for the assessment: Pain: Overall, how severe was your psoriasis-related pain over the past 24 hours?; Itching: Overall, how severe was your psoriasis-related itch over the past 24 hours?; & Scaling: Overall, how severe was your psoriasis related scaling over the past 24 hours? Patients had to rate their pain, itching, & scaling from 0 to 10 (11-point scale), with the understanding that the 0 represents the absence or null end of the pain, itching, or scale intensity (i.e. no pain, itching or scaling) & the 10 represents the other extreme of pain, itching, or scaling intensity (i.e. pain, itching or scaling as bad as it could be). The number that the patient selected represents his or her intensity score in the respective category.
Time Frame: 16 and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
Number analyzed (Participants) | 662 | 673 | 324 | 1659
scores on a scale
  Pain: Wk 16: number analyzed (Participants) | 640 | 649 | 310 | 1599
  Pain: Wk 16 | -3.0 (2.87) | -3.3 (3.11) | -3.3 (3.30) | -3.2 (3.06)
  Pain: Wk 52: number analyzed (Participants) | 645 | 657 | 316 | 1618
  Pain: Wk 52 | -3.1 (2.95) | -3.2 (3.22) | -3.3 (3.36) | -3.2 (3.14)
  Itching: Wk 16: number analyzed (Participants) | 640 | 649 | 311 | 1600
  Itching: Wk 16 | -4.9 (2.96) | -4.9 (3.06) | -4.8 (3.31) | -4.9 (3.07)
  Itching: Wk 52: number analyzed (Participants) | 646 | 656 | 317 | 1619
  Itching: Wk 52 | -5.0 (2.92) | -5.0 (3.10) | -4.6 (3.28) | -4.9 (3.07)
  Scaling: Wk 16: number analyzed (Participants) | 640 | 650 | 312 | 1602
  Scaling: Wk 16 | -5.5 (2.68) | -5.5 (2.71) | -5.2 (3.26) | -5.4 (2.81)
  Scaling: Wk 52: number analyzed (Participants) | 646 | 657 | 317 | 1620
  Scaling: Wk 52 | -5.4 (2.72) | -5.3 (2.87) | -4.9 (3.27) | -5.3 (2.90)

9. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Scale Scores at Week 16 and Week 52
Description: Treatment Satisfaction Questionnaire for Medication (TSQM) is general measure for treatment satisfaction. Each scale score was calculated by summing individual items and then transformed to a 0-100 scale. Higher summary scores indicate better satisfaction with study drug.
Time Frame: 16 and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
Number analyzed (Participants) | 662 | 673 | 324 | 1659
scores on a scale
  Effectiveness: Wk 16: number analyzed (Participants) | 650 | 668 | 318 | 1636
  Effectiveness: Wk 16 | 81.5 (24.02) | 80.9 (25.13) | 75.0 (23.43) | 80.0 (24.48)
  Effectiveness: Wk 52: number analyzed (Participants) | 655 | 671 | 322 | 1648
  Effectiveness: Wk 52 | 85.1 (20.64) | 82.0 (25.05) | 74.9 (24.24) | 81.9 (23.50)
  Convenience: Wk 16: number analyzed (Participants) | 650 | 668 | 319 | 1637
  Convenience: Wk 16 | 79.2 (15.50) | 80.8 (15.83) | 75.9 (15.20) | 79.2 (15.67)
  Convenience: Wk 52: number analyzed (Participants) | 655 | 671 | 323 | 1649
  Convenience: Wk 52 | 82.8 (15.67) | 83.9 (15.42) | 78.9 (15.14) | 82.5 (15.57)
  Global satisfaction: Wk 16: number analyzed (Participants) | 650 | 668 | 319 | 1637
  Global satisfaction: Wk 16 | 83.8 (14.71) | 83.3 (16.68) | 75.1 (20.07) | 81.9 (16.99)
  Global satisfaction: Wk 52: number analyzed (Participants) | 655 | 671 | 322 | 1648
  Global satisfaction: Wk 52 | 83.9 (17.23) | 81.9 (20.38) | 73.5 (23.10) | 81.1 (20.14)

10. Secondary Outcome: Patient Benefit Index (PBI) at Week 16 and Week 52
Description: The questionnaire includes 23 items on patient-relevant therapy needs & benefits. The first part of the instrument, the 'Patient Needs Questionnaire' (PNQ), is filled in by the patient before therapy. A 5-step Likert scale (0='not important at all' to 4='very important') records the individual relevance of the different items to the patients. The second part, the PBQ, is filled in by the patient during or after therapy. It comprises the same items as the PNQ, but in contrast, the patients evaluate the extent to which the treatment needs have been fulfilled by therapy (scaled from 0='treatment did not help at all' to 4='treatment helped a lot'). In addition, the Likert scale contains the option 'does not apply to me' in the PNQ & the option 'did not apply to me' in the PBQ. The needs prior to treatment (PNQ) & the benefits achieved by treatment (PBQ) are converted to a weighted index value, the PBI in the narrower sense. PBI can have a value from 0='no benefit' to 4='maximal benefit'.
Time Frame: Week 16 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
Number analyzed (Participants) | 662 | 673 | 324 | 1659
scores on a scale
  Week 16: number analyzed (Participants) | 439 | 472 | 226 | 1137
  Week 16 | 3.5 (0.61) | 3.4 (0.69) | 3.2 (0.85) | 3.4 (0.70)
  Week 52: number analyzed (Participants) | 509 | 532 | 253 | 1294
  Week 52 | 3.5 (0.70) | 3.4 (0.80) | 3.2 (0.96) | 3.4 (0.80)

ADVERSE EVENTS:
Time Frame: All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit for up to 52 weeks.
Arm/Group | Subpopulation A (Naive) | Subpopulation B (Non-biologic) | Subpopulation C (Biologic) | All Participants
All-Cause Mortality (participants affected / at risk) | 0/663 | 0/673 | 1/324 | 1/1660
Serious Adverse Events (participants affected / at risk) | 43/663 | 44/673 | 32/324 | 119/1660
Other Adverse Events (participants affected / at risk) | 450/663 | 474/673 | 203/324 | 1127/1660
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subpopulation A (Naive) (N=663) | Subpopulation B (Non-biologic) (N=673) | Subpopulation C (Biologic) (N=324) | All Participants (N=1660)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2 | 0 | 4
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 1
Pupils unequal (Eye disorders) | 0 | 0 | 1 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 3 | 0 | 4
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 2
Sudden death (General disorders) | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 1
Dermo-hypodermitis (Infections and infestations) | 0 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 4 | 2 | 0 | 6
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 1
Otitis media chronic (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Purulent discharge (Infections and infestations) | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Type 3 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 1
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 | 0 | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 3 | 3
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 2
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 2 | 3
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 5
Hypertension (Vascular disorders) | 2 | 0 | 0 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subpopulation A (Naive) (N=663) | Subpopulation B (Non-biologic) (N=673) | Subpopulation C (Biologic) (N=324) | All Participants (N=1660)
Diarrhoea (Gastrointestinal disorders) | 35 | 30 | 14 | 79
Toothache (Gastrointestinal disorders) | 14 | 15 | 5 | 34
Asthenia (General disorders) | 16 | 10 | 7 | 33
Fatigue (General disorders) | 17 | 25 | 6 | 48
Influenza like illness (General disorders) | 8 | 15 | 4 | 27
Pyrexia (General disorders) | 11 | 12 | 8 | 31
Bronchitis (Infections and infestations) | 24 | 27 | 10 | 61
Conjunctivitis (Infections and infestations) | 33 | 21 | 15 | 69
Folliculitis (Infections and infestations) | 16 | 21 | 7 | 44
Gastroenteritis (Infections and infestations) | 21 | 14 | 6 | 41
Influenza (Infections and infestations) | 15 | 17 | 8 | 40
Nasopharyngitis (Infections and infestations) | 189 | 189 | 66 | 444
Oral candidiasis (Infections and infestations) | 16 | 30 | 14 | 60
Oral herpes (Infections and infestations) | 16 | 8 | 7 | 31
Otitis externa (Infections and infestations) | 9 | 7 | 7 | 23
Pharyngitis (Infections and infestations) | 28 | 19 | 10 | 57
Rhinitis (Infections and infestations) | 37 | 37 | 11 | 85
Sinusitis (Infections and infestations) | 11 | 16 | 11 | 38
Tinea pedis (Infections and infestations) | 16 | 18 | 7 | 41
Tonsillitis (Infections and infestations) | 22 | 34 | 11 | 67
Upper respiratory tract infection (Infections and infestations) | 39 | 25 | 20 | 84
Urinary tract infection (Infections and infestations) | 26 | 21 | 13 | 60
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 28 | 18 | 72
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 46 | 15 | 92
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 7 | 7 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 17 | 7 | 39
Tendonitis (Musculoskeletal and connective tissue disorders) | 6 | 1 | 7 | 14
Headache (Nervous system disorders) | 76 | 79 | 21 | 176
Haematuria (Renal and urinary disorders) | 10 | 17 | 5 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 31 | 12 | 80
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 34 | 40 | 14 | 88
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 7 | 8 | 18
Eczema (Skin and subcutaneous tissue disorders) | 25 | 20 | 5 | 50
Intertrigo (Skin and subcutaneous tissue disorders) | 12 | 15 | 3 | 30
Pruritus (Skin and subcutaneous tissue disorders) | 31 | 41 | 13 | 85
Psoriasis (Skin and subcutaneous tissue disorders) | 20 | 36 | 22 | 78
Urticaria (Skin and subcutaneous tissue disorders) | 14 | 7 | 3 | 24
Hypertension (Vascular disorders) | 26 | 31 | 8 | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT02752776/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT02752776/SAP_001.pdf